CLINICAL TRIAL: NCT06027385
Title: Scientific Basis for a Newborn Screening for Cystinosis and Spinal Muscular Atrophy
Brief Title: Genetic Newborn Screening for Cystinosis and Spinal Muscular Atrophy
Acronym: GENESIS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cystinose Stiftung (Other)
Collaborators: Labor Becker & Kollegen, Munich, Germany (Unknown); Screening Labor Hannover (Other); Genetikum, Ulm, Germany (Unknown); Bavarian State Office of Health and Food Safety (LGL), Unterschleißheim, Germany (Unknown); Internal Medicine, Freiburg University Hospital, Freiburg, Germany (Unknown); Attorney DSZ Rechtsanwälte GmbH, Barkhovenallee 1, 45239 Essen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017-GEN1
Record Dates: First submitted 2023-08-17; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Cystinosis; Cystinosis, Nephropathic; Spinal Muscular Atrophy
Keywords: Newborn Screening; Screening; Molecular-based Screening
MeSH Terms: conditions — Cystinosis; Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: All newborns whose parents have agreed to participate in the pilot project will be tested for three mutations in the CTNS gene and a homozygous deletion of exon 7 in the SMN1-gene.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tested Newborns (Experimental): Tested for three mutations in the CTNS gene and one mutation in the SMN1 gene.
  Interventions: Diagnostic Test: molecular-based screening

INTERVENTIONS:
Diagnostic Test: molecular-based screening — Test for three mutations in the CTNS gene and one mutation in the SMA1 gene.

SUMMARY:
Newborn screening in Germany is a voluntary program. Cystinosis and spinal muscular atrophy (SMA) are rare autosomal recessive diseases. They are inherited in an autosomal recessive manner, i.e. both parents carry a defective gene. Neither disease can be detected early by the methods established in routine newborn screening. However, common genetic mutations are known for both diseases.

The aim of the study presented here is to provide the scientific basis for molecular genetic newborn screening for cystinosis and SMA. In particular, to investigate whether inclusion of these diseases in general newborn screening should be recommended.

The participating screening laboratories for this project are Labor Becker & Kollegen, Munich, Germany and Screening Laboratory Hannover, Germany. Hospitals that send their dry blood spot cards for routine newborn screening to these laboratories will receive an offer to participate in the pilot project. Participation is free of charge.

Parents who wish to participate in this pilot project will receive an information sheet explaining the screening process and objectives. A parent and the treating physician sign the information sheet as documentation of informed consent. Their signature and informed consent are required for the pilot.

Routine NBS according to German pediatric guidelines involves the collection of dried blood spot cards 36-72 hours after birth. Molecular genetic screening in the pilot project will be performed with the same dried blood spot card used for routine newborn screening.

In cystinosis, genetic testing for the 3 most common mutations in Germany will be performed. In SMA, a homozygous deletion of exon 7 in the SMN gene is detected by a PCR test. The molecular genetic test is performed on the same day as routine newborn screening.Normal findings are not reported to parents. However, they can contact the laboratories to inquire about them.

Parents of newborns with two mutations in the cystinosis gene or with a homozygous deletion of exon 7 in the SMN gene are immediately informed of the disease by a physician. Further diagnostics to confirm the disease will be organized close to home.

The study started on Jan. 15, 2018, and recruitment was completed on Sept. 30, 2022.

DETAILED DESCRIPTION:
Population-based newborn screening (NBS) is an important public health program that has vastly improved the course of several diseases through early detection. The selection of screened disorders generally follows the 10 principles outlined by Wilson and Jungner. In Germany, NBS has been a voluntary National Health Service program since 1969 which currently covers 17 disorders. Current NBS methods, which employ tandem mass-spectrometric analysis of newborn dried blood spots, cannot detect many potentially treatable genetic conditions. At the same time, molecular-based NBS is increasingly feasible because DNA can be extracted from a dried blood spot, next generation sequencing has become economical, and molecular diagnostics have greater reliability and increased validity as genetic databases become more refined and comprehensive. Nephropathic cystinosis and spinal muscular atrophy (SMA) are eligible for molecular-based NBS because effective therapies are available.

This study will provide a scientific basis for newborn screening for cystinosis and SMA and investigate whether inclusion of these diseases in general newborn screening should be recommended. By observing identified infants compared to symptomatically diagnosed patients outside the pilot project, we will determine whether and to what extent early diagnosis and initiation of therapy leads to a more favorable prognosis.

Cystinosis: Cystinosis is a rare autosomal recessive systemic disease with high morbidity and mortality caused by pathogenic variants in the CTNS gene that encodes the lysosomal cystine transporter cystinosin, leading to accumulation of cystine within the lysosome. Life-long cystine-depleting therapy with oral cysteamine, the only specific therapy for cystinosis, along with the availability of renal replacement therapy in childhood, has dramatically improved patient outcomes. There is robust evidence that early initiation and sustained therapy with cysteamine are both essential for delaying progression to chronic kidney disease (CKD) and end-organ damage.

Currently, the diagnosis of cystinosis is based on the presence of elevated cystine levels in white blood cells. This method is unsuitable for NBS.

Spinal Muscular Atrophy (SMA): Spinal muscular atrophy has a prevalence of approximately 1:10,000 live births in Germany. It is inherited in an autosomal recessive manner. Newborns with spinal muscular atrophy are without clinical symptoms after birth.

The cause of spinal muscular atrophy is a deletion of exon 7 in the SMN1 gene, the coding gene for the "survival motor neuron protein". Homozygous deletion lacks the functional SMN protein on which the anterior horn cells in the spinal cord depend. Heterozygous carriers are asymptomatic. Lack of the functional SMN protein results in damage to motor neurons at the spinal cord level, leading to severe neurogenic remodeling and atrophy of skeletal muscles.

In addition to the SMN1 gene, humans have an almost identical, adjacently located "pseudo-gene," the SMN2 gene. It differs from the SMN1 gene only by 5 single base pairs. The SMN2 protein plays no role in healthy humans, since sufficient functional SMN1 protein is present. The SMN2 gene contains a molecular switch that can completely shut down the expression of the gene. The clinical variability of spinal muscular atrophy is explained by differential expression of the SMN2 protein. Thus, the readout of the SMN2 gene including its exon 7 by inhibition of the off switch represents a therapeutic target for the treatment of SMA patients. The possibility of a therapy to positively influence the course of the disease was demonstrated in the placebo-controlled multi-center study with an antisense oligonucleotide nusinersen (Spinraza®) from Ionis/Biogen in 2015/2016.

Diagnosis of the disease in cases of clinical suspicion has been made by targeted testing of the SMN1 and SMN2 genes from EDTA blood and DNA isolated therefrom. The test is usually performed in genetics laboratories using MLPA (multiplex ligation-dependent probe amplification). Because a commercial kit is required for each sample, the test is too costly for screening as part of newborn screening.

Procedure:

Study population Hospitals in Germany are free to choose which of the 11 certified laboratories they send the dry blood spot cards to for newborn screening and whether they want to participate in pilot projects.

In this project, the Becker & Kollegen laboratory in Munich and the Hannover screening laboratory are informing their senders about the possibility of adding genetic screening for cystinosis (Hannover) or cystinosis and SMA (Munich) to the routinely established newborn screening.

The study population includes newborns whose parents wish to participate in the pilot project and have provided written informed consent. An additional information and consent sheet for cystinosis and SMA screening is provided, which includes an explanation of the screening process and objectives, expected benefits, possible adverse consequences of non-participation, and the significance of the test results. Parents are informed that they will be informed of normal, unremarkable results only upon request. Consent must be documented with the signature of at least one parent and the signature of the informing physician on the consent form. The consent form for the pilot project also includes consent to share contact information and findings with a specialized center in the event of an abnormal screening result.

In the event of a positive result, the laboratory must first inform the sender and clarify whether or not the child is still in hospital. If the child is still undergoing inpatient treatment, the sender obtains the initial information from the parents and notifies an expert for the corresponding diagnosis. If the child has already been discharged from the hospital, the laboratory contacts the appropriate expert directly (Cystinosis: Priv.-Doz. Dr. med. Katharina Hohenfellner, Rosenheim; SMA: Prof. Dr. med. Wolfgang Müller-Felber, Munich).

Sampling Molecular genetic screening is performed using the same dry blood card (drops of blood on a filter paper card) as routine NBS. No additional blood collection is required. If little material is available, the regular NBS is performed first, followed by screening for cystinosis and SMA. According to the pediatric guideline, the blood sample for the NBS should be collected between 36 and 72 hours of life.

In general, for all invalid results (i.e., if the control reaction fails) and for all abnormal results the test is repeated internally for confirmation using the available blood sample. If the quality of the blood sample is poor (e.g., too little blood), the laboratory will request a new blood sample. If there is too little material to perform the required next generation sequencing, the laboratory will also request another dried blood sample.

Measurements and Methods Cystinosis: For cystinosis screening, multiplex PCR was performed at the first stage to detect the three most common CTNS mutations in Germany, i.e. a 57kb deletion (responsible for about half of cystinosis in Europe and North America) c.18_21delGACT, p.T7Ffs*7 and c.926dupG, p.S310Qfs*55 . Heterozygous samples will be subjected to amplicon-based next-generation sequencing for 101 pathogenic mutations. This approach predicts a detection rate of 96.5%.

SMA The triplex PCR for the CTNS mutations described above is complemented by another PCR that detects exon 7 in the SMN1 gene. With this quadruplex PCR, a specific signal is obtained for normal samples (those without or with heterozygous exon 7 deletion in both alleles of the SMN1 gene). SMA screening is considered positive if a homozygous exon 7 deletion is detected in the SMN1 gene. The absence of PCR amplification indicates the absence of a functional SMN1 copy, i.e., an affected newborn. Heterozygous individuals cannot be detected by this method Detection rate, false positive and false negative results An overall detection rate of more than 95% is assumed for both diseases. False negative screening results are unlikely. In cystinosis, false negative results are possible due to previously unknown rare mutations or patients not carrying any of the three most common mutations. In SMA, patients in whom a heterozygous deletion is combined with a point mutation are not considered. In patients with symptoms of cystinosis or SMA, further diagnostic tests are performed independently of screening.

False positive screening results are also very unlikely. In cystinosis, a heterozygous sample may falsely appear as homozygous due to "allelic dropout" (PCR failure of an allele due to mutations in the primer binding region).

Confirmation of diagnosis Cystinosis: In patients found to have either a homozygous or compound heterozygous mutation in a CTNS gene, the diagnosis is confirmed by determining the intraleukocytic cystine level from EDTA blood. This sample is sent to the metabolic laboratory in Münster within the first 14 days of life.

SMA: If exon 7 in the SMN1 gene is homozygous, SMA must be assumed (> 50% type I with most severe course). In order to classify the severity of SMA, further diagnostics are required by recording the number of SMN-2 copies. Another blood sample will be sent by the responsible care center to the reference laboratory in Ulm. The verification test results are forwarded to the screening laboratory for quality control.

Care of the affected child Cystinosis: Children with positive cystinosis screening results are referred to the nearest metabolic disease center. Therapy with cysteamine will be started immediately after the diagnosis is confirmed..

SMA: Children with positive SMA screening results are referred either to the Center for Neuromuscular Diseases in the Social Pediatric Center of the Dr. von Hauner Children's Hospital (Bavaria) or to the University Hospitals of Essen and Münster.

Project scope The project was initially limited to 200,000 samples, with the possibility of expansion.

ELIGIBILITY:
Inclusion Criteria:

* Newborns whose dry bloodspot card was sent to screening labs involved in the project
* Consent of guardians

Exclusion Criteria:

* no consent of guardians

Ages: 36 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300000 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with confirmed diagnosis of Cystinosis | up to 60 months
  Newborns identified with 57-kb CTNS mutation homozygous, compound heterozygous , with c.18_21delGACT p.T7Ffs*7 homozygous or compound heterozygous or c.926_927insG, p.S310Qfs * 55 homozygous or compound heterozygous and elevated white blood cell cystine level.
Number of participants with heterozygous mutations | up to 4 weeks
  Newborns identified with heterozygous CTNS mutations of 57-kb CTNS and heterozygous c.18_21delGACT p.T7Ffs*7 mutations and heterozygous c.926_927insG, p.S310Qfs * 55 mutations
Number of participants with confirmed diagnosis of SMA | up to 48 months
  Newborns identified with homozygous deletion of exon 7 in the SMN1-gene
time interval until start of treatment for both diseases | up to 4 weeks
  For both diseases the time interval will be evaluated from the time of identification in screening to the introduction of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Hohenfellner, PD Dr., Study Chair — RoMed Hospital
Locations (4):
- Germany (4):
  - RoMed Hospital, Rosenheim, Bavaria
  - University Hospital Essen, Center for Pediatrics and Adolescent Medicine, Essen
  - Dr. von Haunersches Kinderspital, München
  - University Hospital Münster, Clinic and Polyclinic for Pediatrics and Adolescent Medicine, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hohenfellner K, Elenberg E, Ariceta G, Nesterova G, Soliman NA, Topaloglu R. Newborn Screening: Review of its Impact for Cystinosis. Cells. 2022 Mar 25;11(7):1109. doi: 10.3390/cells11071109. PMID 35406673
- [Background] Vill K, Blaschek A, Schara U, Kolbel H, Hohenfellner K, Harms E, Olgemoller B, Walter MC, Muller-Felber W. [Spinal muscular atrophy : Time for newborn screening?]. Nervenarzt. 2017 Dec;88(12):1358-1366. doi: 10.1007/s00115-017-0447-3. German. PMID 29101527
- [Background] Hohenfellner K, Bergmann C, Fleige T, Janzen N, Burggraf S, Olgemoller B, Gahl WA, Czibere L, Froschauer S, Roschinger W, Vill K, Harms E, Nennstiel U. Molecular based newborn screening in Germany: Follow-up for cystinosis. Mol Genet Metab Rep. 2019 Sep 18;21:100514. doi: 10.1016/j.ymgmr.2019.100514. eCollection 2019 Dec. PMID 31641587
- [Background] Fleige T, Burggraf S, Czibere L, Haring J, Gluck B, Keitel LM, Landt O, Harms E, Hohenfellner K, Durner J, Roschinger W, Becker M. Next generation sequencing as second-tier test in high-throughput newborn screening for nephropathic cystinosis. Eur J Hum Genet. 2020 Feb;28(2):193-201. doi: 10.1038/s41431-019-0521-3. Epub 2019 Sep 30. PMID 31570786
- [Background] Vill K, Kolbel H, Schwartz O, Blaschek A, Olgemoller B, Harms E, Burggraf S, Roschinger W, Durner J, Glaser D, Nennstiel U, Wirth B, Schara U, Jensen B, Becker M, Hohenfellner K, Muller-Felber W. One Year of Newborn Screening for SMA - Results of a German Pilot Project. J Neuromuscul Dis. 2019;6(4):503-515. doi: 10.3233/JND-190428. PMID 31594245
- [Background] Czibere L, Burggraf S, Fleige T, Gluck B, Keitel LM, Landt O, Durner J, Roschinger W, Hohenfellner K, Wirth B, Muller-Felber W, Vill K, Becker M. High-throughput genetic newborn screening for spinal muscular atrophy by rapid nucleic acid extraction from dried blood spots and 384-well qPCR. Eur J Hum Genet. 2020 Jan;28(1):23-30. doi: 10.1038/s41431-019-0476-4. Epub 2019 Jul 30. PMID 31363188